CLINICAL TRIAL: NCT02949999
Title: A Single-center, Double-blind, Placebo-controlled, Randomized, Ascending Multiple-dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of Voclosporin in Healthy Japanese Volunteers
Brief Title: Voclosporin in Healthy Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUR-VCS-2015-J01
Record Dates: First submitted 2016-10-20; First posted 2016-10-31 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Volunteers
Keywords: Calcineurin inhibitor; Voclosporin
MeSH Terms: interventions — voclosporin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0.25mg/kg voclosporin (Experimental): 0.25mg/kg voclosporin BID.
  Interventions: Drug: Voclosporin
- 0.5mg/kg voclosporin (Experimental): 0.5mg/kg voclosporin BID
  Interventions: Drug: Voclosporin
- 1.0mg/kg voclosporin (Experimental): 1.0mg/kg voclosporin BID
  Interventions: Drug: Voclosporin
- 1.5mg/kg voclosporin (Experimental): 1.5mg/kg voclosporin BID
  Interventions: Drug: Voclosporin
- Placebo voclosporin (Placebo Comparator): placebo BID
  Interventions: Drug: Voclosporin

INTERVENTIONS:
Drug: Voclosporin
  Other Names: ISA247

SUMMARY:
The study is a single-centre, double-blind, placebo controlled, randomized, ascending multiple dose study to assess the safety, tolerability, pharmacokinetics and pharmacodynamic profiles of voclosporin.

DETAILED DESCRIPTION:
Ten subjects will be randomized into each of four treatment groups to receive approximately 0.25, 0.5, 1.0, 1.5mg/kg/dose of voclosporin vs placebo. For Day 1, subjects will be given oral treatment once a day; Day 2, subjects will not be given any oral treatment; Day 3-12, subjects will be given oral treatment twice a day; Day 13, subjects will be given oral treatment once a day. The duration of the study takes about 21 days (including follow up assessments).

ELIGIBILITY:
Key Inclusion Criteria:

* Japanese males and females by birth aged 20 - 45 years inclusive
* Females who are non-pregnant, non-lactating, and either post-menopausal for at least 1 year, surgically sterile for at least 3 months, or from 35 days prior to study entry (i.e. Day -2) until 30 days following study completion/discharge and using an approved method of contraception.
* Males who are sterile or from the time of dose administration until 30 days following their dose administration and using an approved method of contraception.
* Screening FSH >40 IU/ml in self-identified post-menopausal female subjects.
* Weight must be >55 kg but <100 kg, with BMI of 18-30 kg/m2 inclusive.
* Healthy as defined by normal screening assessments, including full medical history, complete physical examination, vital signs, 12-lead ECG, hematology, blood chemistry and urinalysis. Laboratory results must be within the reference range or considered to be not clinically significant by the Principal Investigator with agreement of the Medical Monitor. Lab tests may be repeated during the screening period as appropriate.
* Capable to participate, provide informed consent and comply with study procedures and restrictions
* Must agree to refrain from consumption of grapefruit juice from at least one week prior to dosing until all follow-up procedures are completed.

Key Exclusion Criteria:

* History of drug abuse and/or alcoholism in the previous 2 years.
* Positive urine drug test, urine cotinine test or alcohol breath test at screening.
* Positive for Hepatitis B, Hepatitis C or HIV.
* QTcB >430 msec in males, or QTcB >450 msec in females in 12-lead ECG tracing at screening.
* Blood donation within 56 days prior to dosing and plasma donation within 7 days prior to first dosing.
* Hemoglobin value < 12 g/dL.
* Current smokers (smoking cigarettes and other forms of tobacco or nicotine use must be stopped at least 90 days before screening).
* History of alcohol consumption averaging more than 2 drinks per day in a week (1 drink is 12 oz beer, 4 oz wine or 1.5oz of spirits) within 6 months prior to screening. Alcohol-containing foods or beverages are prohibited within 7 days prior to study entry and during the entire study duration.
* Use of any drugs known to inhibit or induce hepatic drug metabolism (i.e. inducers include barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; inhibitors include antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to administration of the study medication.
* Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days (90 days for biologics) prior to the first dosing
* Use of prescription medication within 14 days prior to first dosing or over-the-counter products (including natural products, vitamins, garlic as supplement) within 7 days prior to first dosing, except for topical products without systemic absorption, or is likely to need medication during the study period.
* Clinically significant abnormal liver function, abnormal renal function, active tuberculosis (TB), or known history of TB/evidence of old TB if not taking prophylaxis with isoniazid, current or recent infections, history of hypertension and history of malignancy.
* Any reason which, in the opinion of the Principal Investigator or the Sponsor's medical monitor, would prevent the subject from participating in the study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 21 days
  Tolerability of voclosporin after single and multiple oral ascending doses
Mean, median and standard deviation of laboratory parameters. Incidence of laboratory parameters outside of normal range | 21 days
  Safety of voclosporin after single and multiple oral ascending doses

SECONDARY OUTCOMES:
Pharmacokinetics of voclosporin after single and multiple oral ascending doses | 21 days
  Peak Plasma Concentration (Cmax)
Pharmacokinetics of voclosporin after single and multiple oral ascending doses | 21 days
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- MAD VCS Site, Dasmariñas, Cavite, Philippines

IPD SHARING:
Plan to Share IPD: No